CLINICAL TRIAL: NCT04219085
Title: CAPO: Continuous Glucose Monitoring in A2 Gestational Diabetes and Pregnancy Outcomes
Acronym: CAPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2000027143; 000 (Other: CTGTY)
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Results first posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Gestational Diabetes; Maternal Complication of Pregnancy
Keywords: gestational diabetes; fetal or neonatal outcomes; maternal morbidity
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Intervention Model Description: randomized controlled trial, not blinded
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Routine Care (Active Comparator): Monitoring of control of gestational diabetes with routine care and use of a glucometer and fingersticks 4 times a day
  Interventions: Other: Routine Care
- Continuous Glucose Monitor (Experimental): Monitoring of control of gestational diabetes with use of a continuous glucose monitor
  Interventions: Device: Continuous Glucose Monitor

INTERVENTIONS:
Device: Continuous Glucose Monitor — Wearing of a continuous glucose monitor to monitor blood glucose levels in women with gestational diabetes
  Arms: Continuous Glucose Monitor
Other: Routine Care — Use of a glucometer to monitor blood glucose levels in women with gestational diabetes
  Arms: Routine Care

SUMMARY:
This study will utilize continuous glucose monitoring in women with A2 gestational diabetes. Women will be randomized to continuous glucose monitoring or routine care with fingersticks to check their blood glucose four times daily. It is hypothesized that women in the continuous glucose monitoring arm will have a lower incidence of the composite primary outcome, which includes the following variables: perinatal death, shoulder dystocia, birth weight greater than 4,000 grams, NICU admission for treatment of hypoglycemia (blood glucose level <40mg/dL) and birth trauma, including fracture or nerve palsy.

DETAILED DESCRIPTION:
Diabetes complicates 6-7% of pregnancies annually and approximately 85% of these cases are women diagnosed with gestational diabetes (GDM).1,2 The prevalence of GDM varies within populations based on obesity rates, maternal age and ethnicity. GDM is diagnosed during the third trimester through a two-step process of a 50-gram oral glucose challenge screen and a subsequent 100-gram oral glucose challenge test if the woman screens positive. Once the diagnosis is confirmed women are asked to monitor their glucose levels with finger sticks at least four times a day (fasting and post-prandial) and medication is added when glucose target goals cannot be reached by diet and exercise alone. Approximately, 15% of women will not reach glucose target goals with diet and exercise alone and will require medication. These women are then diagnosed with class A2 GDM by the White classification of diabetes.

Identification of women with GDM who require treatment is essential in optimizing pregnancy outcomes for these women. Treatment of GDM results in lower neonatal morbidity, reduced incidence of large for gestational age infants (LGA), reduced incidence of preeclampsia and shoulder dystocia and a reduced need for cesarean delivery.3-5 Since LGA infants are at higher risk for hypoglycemia which may necessitate admission to the neonatal intensive care unit (NICU), treatment of GDM reduces the incidence of LGA infants resulting in less hypoglycemia and NICU admissions.

Given that pregnancy outcomes are directly tied to blood glucose control, it is essential that women with GDM play an active role in the monitoring of their disease. The frequency of monitoring and frustration with diet can lead to issues with patient compliance and ultimately impact their pregnancy outcomes. One study found that just over half of women successfully tested their blood glucose via finger sticks ≥ 80% of the time. About 25% of the women in the same study had <90% of the values matching in their glucometer and their blood glucose log.6 Given these issues with compliance the need for a better and more convenient monitoring system is evident. Continuous glucose monitors (CGM) are a relatively new device that have yet to be fully explored for their utility in pregnancy. The current generation of CGM has had exponential growth in the clinical care of diabetes, driven primarily by the improved accuracy of these devices, longer duration sensor life (ranging from 7-14 days in currently available models), and the ability to collect these data without performing calibration of the sensors with fingerstick glucose readings. Continuous Glucose Monitoring in Women with Type 1 Diabetes in Pregnancy Trial (CONCEPTT), demonstrated the utility of CGM data to decrease the frequency of adverse neonatal outcomes in a pregestational diabetes population.7 A more recent trial of blinded CGM data in women with GDM showed mean sensor glucose was significantly higher in women who delivered LGA infants. The 24-hour mean glucose was different between groups in this study (112 mg/dL vs. 104 mg/dL, p=0.025), driven by higher overnight mean glucose levels (108 mg/dL vs. 99 mg/dL, p=0.005).8 Given that this is not a time that women with GDM would normally be monitoring their blood sugar it is evident that CGM may be useful, not only in increasing patient compliance by eliminating the need for measuring serum glucose via finger sticks and a glucometer four times a day but by allowing for monitoring of blood glucose levels at times that are not normally convenient for testing.

ELIGIBILITY:
Inclusion Criteria:

* women between 18-50 years old
* pregnant
* singleton gestation
* diagnosis of gestational diabetes requiring medication (A2) during the current pregnancy between 24-36 weeks' gestation

Exclusion Criteria:

* pregestational diabetes
* diagnosis with gestational diabetes < 24 weeks gestation or > 36 weeks gestation
* known fetal anomalies
* fetal growth restriction diagnosed during the current pregnancy
* diagnosis of polyhydramnios at time of randomization
* abnormal diagnostic genetic testing or genetic screening for the fetus in the current pregnancy prior to randomization
* twin or higher order multiple gestation
* non-compliance with prenatal visits (missing ≥3 visits prior to enrollment) prior to diagnosis with A2 gestational diabetes
* maternal medical comorbidities including the following: lupus, chronic hypertension, cancer, ischemic cardiovascular disease

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — ongoing pregnancy is required for study
Enrollment: 65 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Merriam, MD, MS, Principal Investigator — Assistant Professor; Assistant Professor, Department of Obstetrics, Gynecology and Reproductive Sciences
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No
no plan to share

REFERENCES:
- [Background] Martin JA, Hamilton BE, Osterman MJK, Driscoll AK, Drake P. Births: Final Data for 2017. Natl Vital Stat Rep. 2018 Nov;67(8):1-50. PMID 30707672
- [Background] The American College of Obstetricians and Gynecologists Practice Bulletin Number 190. Gestational Diabetes Mellitus. February 2018.
- [Background] Crowther CA, Hiller JE, Moss JR, McPhee AJ, Jeffries WS, Robinson JS; Australian Carbohydrate Intolerance Study in Pregnant Women (ACHOIS) Trial Group. Effect of treatment of gestational diabetes mellitus on pregnancy outcomes. N Engl J Med. 2005 Jun 16;352(24):2477-86. doi: 10.1056/NEJMoa042973. Epub 2005 Jun 12. PMID 15951574
- [Background] Landon MB, Spong CY, Thom E, Carpenter MW, Ramin SM, Casey B, Wapner RJ, Varner MW, Rouse DJ, Thorp JM Jr, Sciscione A, Catalano P, Harper M, Saade G, Lain KY, Sorokin Y, Peaceman AM, Tolosa JE, Anderson GB; Eunice Kennedy Shriver National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. A multicenter, randomized trial of treatment for mild gestational diabetes. N Engl J Med. 2009 Oct 1;361(14):1339-48. doi: 10.1056/NEJMoa0902430. PMID 19797280
- [Background] Hartling L, Dryden DM, Guthrie A, Muise M, Vandermeer B, Donovan L. Benefits and harms of treating gestational diabetes mellitus: a systematic review and meta-analysis for the U.S. Preventive Services Task Force and the National Institutes of Health Office of Medical Applications of Research. Ann Intern Med. 2013 Jul 16;159(2):123-9. doi: 10.7326/0003-4819-159-2-201307160-00661. PMID 23712381
- [Background] Cosson E, Baz B, Gary F, Pharisien I, Nguyen MT, Sandre-Banon D, Jaber Y, Cussac-Pillegand C, Banu I, Carbillon L, Valensi P. Poor Reliability and Poor Adherence to Self-Monitoring of Blood Glucose Are Common in Women With Gestational Diabetes Mellitus and May Be Associated With Poor Pregnancy Outcomes. Diabetes Care. 2017 Sep;40(9):1181-1186. doi: 10.2337/dc17-0369. Epub 2017 Jul 19. PMID 28724718
- [Background] Law GR, Alnaji A, Alrefaii L, Endersby D, Cartland SJ, Gilbey SG, Jennings PE, Murphy HR, Scott EM. Response to Comment on Law et al. Suboptimal Nocturnal Glucose Control Is Associated With Large for Gestational Age in Treated Gestational Diabetes Mellitus. Diabetes Care 2019;42:810-815. Diabetes Care. 2019 Jul;42(7):e123-e124. doi: 10.2337/dci19-0018. No abstract available. PMID 31221709
- [Background] Feig DS, Donovan LE, Corcoy R, Murphy KE, Amiel SA, Hunt KF, Asztalos E, Barrett JFR, Sanchez JJ, de Leiva A, Hod M, Jovanovic L, Keely E, McManus R, Hutton EK, Meek CL, Stewart ZA, Wysocki T, O'Brien R, Ruedy K, Kollman C, Tomlinson G, Murphy HR; CONCEPTT Collaborative Group. Continuous glucose monitoring in pregnant women with type 1 diabetes (CONCEPTT): a multicentre international randomised controlled trial. Lancet. 2017 Nov 25;390(10110):2347-2359. doi: 10.1016/S0140-6736(17)32400-5. Epub 2017 Sep 15. PMID 28923465

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Routine Care | Continuous Glucose Monitor
Started | 30 | 35
Completed | 30 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Routine Care | Continuous Glucose Monitor | Total
Number analyzed (Participants) | 30 | 35 | 65
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 35 | 65
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 35 | 65
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 11
  Not Hispanic or Latino | 23 | 31 | 54
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 5 | 9
  White | 20 | 22 | 42
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 30 | 35 | 65
Gravidity [Count of Participants; unit: Participants] — Number of prior pregnancies
  Participants
    1 pregnancy | 9 | 6 | 15
    2 pregnancies | 11 | 10 | 21
    ≥3 pregnancies | 10 | 19 | 29
Living Children [Number; unit: participants] — Number of participants with living children
  participants
    0 children | 14 | 12 | 26
    1child | 9 | 13 | 22
    ≥2 children | 7 | 10 | 26
Participant Body Mass Index (BMI) at Delivery [Count of Participants; unit: Participants]
  <25 kg/m^2 | 0 | 2 | 2
  25-<30 kg/m^2 | 2 | 4 | 6
  30-<35 kg/m^2 | 5 | 10 | 15
  35-<40 kg/m^2 | 10 | 9 | 19
  ≥40 kg/m^2 | 13 | 10 | 23
Insurance Type [Count of Participants; unit: Participants]
  Medicaid | 5 | 9 | 14
  Private | 25 | 26 | 51
Medication Type [Count of Participants; unit: Participants] — Type of medication participant was taking at time of enrollment.
  Participants
    Insulin | 29 | 35 | 64
    Metformin | 2 | 0 | 2
History of Gestational Diabetes Mellitus (GDM) [Count of Participants; unit: Participants] | 9 | 5 | 14
Family History of GDM [Count of Participants; unit: Participants] | 13 | 13 | 26
Gestational Age at GDM diagnosis [Mean (Standard Deviation); unit: weeks] | 24.5 (1.1) | 26 (28.2) | 25.3 (5.7)
Gestational Age Starting Medications for GDM [Mean (Standard Deviation); unit: weeks] | 27.4 (4.6) | 28.2 (5.5) | 27.8 (5.0)
Gestational Age at Delivery [Mean (Standard Deviation); unit: weeks] | 37.7 (1.4) | 38 (1.3) | 37.9 (1.3)

OUTCOME MEASURES:

1. Primary Outcome: Composite Primary Outcome
Description: The number of participants who have at least one of each of the following outcome measures occur: perinatal death, shoulder dystocia, birth weight less than 4,000 grams, NICU admission for treatment of hypoglycemia (blood glucose level <40mg/dL) and birth trauma, including fracture or nerve palsy. Any one of these would make the composite primary outcome positive and will be recorded as a categorical variable.
Time Frame: from enrollment up until delivery by 41 weeks gestation, up to 19 weeks total
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Care | Continuous Glucose Monitor
Number analyzed (Participants) | 30 | 35
Participants
  Perinatal Death | 0 | 0
  Shoulder Dystocia | 0 | 0
  Birthweight < 4,000 grams | 4 | 6
  NICU Admission for Hypoglycemia | 4 | 4
  Birth Trauma | 0 | 0
Statistical Analysis 1: Comparison: Routine Care vs Continuous Glucose Monitor; Test type: Superiority; p = 1.0, t-test, 2 sided

2. Secondary Outcome: Cesarean Delivery for an Arrest of Labor Disorder
Description: The number of women who undergo a cesarean delivery for arrest of dilation or descent during labor or induction of labor. This will be recorded as a categorical (yes/no) variable. Data presented below is for the participants that had c-section for arrest.
Time Frame: during delivery by 40 weeks gestation
Population: Out of women who had c-sections
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Care | Continuous Glucose Monitor
Number analyzed (Participants) | 22 | 15
Participants | 1 | 4
Statistical Analysis 1: Comparison: Routine Care vs Continuous Glucose Monitor; Test type: Superiority; p = 0.03, t-test, 2 sided

3. Secondary Outcome: Hypertensive Disorders of Pregnancy.
Description: The number of women who receive a diagnosis of a hypertensive disorder of pregnancy (gestational hypertension, preeclampsia, HELLP). This will be recorded as a categorical (yes/no) variable
Time Frame: from enrollment, through delivery by 41 weeks gestation and the immediate postpartum hospitalization up to 7 days postpartum, up to 20 weeks total
Measure: Count of Participants; unit: Participants
Arm/Group | Routine Care | Continuous Glucose Monitor
Number analyzed (Participants) | 30 | 35
Participants | 5 | 7
Statistical Analysis 1: Comparison: Routine Care vs Continuous Glucose Monitor; Test type: Superiority; p = 0.85, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: from enrollment to 7 days post partum, up to 20 weeks total
Arm/Group | Routine Care | Continuous Glucose Monitor
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/35
Other Adverse Events (participants affected / at risk) | 0/30 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-11-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT04219085/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/85/NCT04219085/ICF_001.pdf